CLINICAL TRIAL: NCT03534037
Title: The Cardiovascular Effects of Febuxostat and Benzbromarone on Left Ventricle Diastolic Dysfunction in Individuals With Metabolic Syndrome and Hyperuricemia - an Open-label Non-blinded Randomized-controlled Clinical Trial
Brief Title: Urate Lowering Therapies and Left Ventricular Diastolic Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Cheng-Wei Liu, Principal investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-107-05-112
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hyperuricemia; Metabolic Syndrome; Left Ventricular Diastolic Dysfunction
Keywords: Serum uric acid; Metabolic syndrome; Left ventricular diastolic dysfunction; Febuxostat; Benzbromarone
MeSH Terms: conditions — Hyperuricemia; Metabolic Syndrome; Ventricular Dysfunction, Left | interventions — Febuxostat; Benzbromarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Febuxostat 40mg (Experimental): Febuxostat 40mg orally per day
  Interventions: Drug: Febuxostat 40 mg
- Benzbromarone 50mg (Active Comparator): Benzbromarone 50mg orally per day
  Interventions: Drug: Benzbromarone 50mg
- Control (Other): Dietary control only
  Interventions: Other: Control

INTERVENTIONS:
Drug: Febuxostat 40 mg — Febuxostat 40 mg orally per day plus dietary control only
  Other Names: Feburic
  Arms: Febuxostat 40mg
Drug: Benzbromarone 50mg — Benzbromarone 50mg orally per day plus dietary control only
  Other Names: Nogout
  Arms: Benzbromarone 50mg
Other: Control — Dietary control only
  Arms: Control

SUMMARY:
Hyperuricemia is an additional risk factor for cardiovascular disease, associating with left ventricular diastolic dysfunction in individuals with metabolic syndrome. The effect of urate-lowering therapies on left ventricular diastolic dysfunction remains unclear. The study is conducted to investigate whether febuxostat or benzbromarone might improve left ventricular diastolic dysfunction in individuals with metabolic syndrome and hyperuricemia

DETAILED DESCRIPTION:
Between 1, July 2018 and 31, Dec 2018, consecutive individuals with metabolic syndrome hyperuricemia are candidates of the present study. After the eligible candidates sign the informed consent, they will receive blood tests with a fasting time of 8 hours at least. The investigators will randomize the study participants by pre-specified random codes with a 1:1:1 ratio to the three groups. The study medication, febuxostat or benzbromarone, will be administered orally on the next day after transthoracic echocardiography is performed. The control group will only receive dietary control. All participant will receive transthoracic echocardiography and blood tests at baseline and at 3 months. The visit will be scheduled at baseline and at the 3rd month. The blood tests include high-sensitivity C-reactive protein, high-sensitivity interleukin-1 beta, high-sensitivity interleukin-6, tumor necrosis factor alpha, Dickkopf-related protein 3, galectin-3, ST2, fibroblast growth factor 23, xanthine oxidase activity, and thioredoxin.

ELIGIBILITY:
Inclusion Criteria (all of the four criteria)

1. Aged between 40-75 years
2. Metabolic syndrome
3. Hyperuricemia, defined as a serum uric acid level of 7 mg/dl or more in men or 6 mg/dl or more in females, with a history of hyperuricemia within a year; or a serum uric acid level of 8 mg/dl or more in men or 7 mg/dl or more in females and it is hardly expected to be modified by dietary control; or persistent hyperuricemia after dietary control for 3 months
4. Not take any of urate-lowering therapies (benzbromarone, allopurinol, or febuxostat)

Exclusion Criteria:

1. pregnancy
2. hypersensitivity to febuxostat or benzbromarone
3. acute gout
4. a history of urinary tract stone
5. chronic kidney disease stage IV or V
6. valvular heart disease with moderate or severe regurgitation
7. left ventricular ejection fraction of 40% or less
8. hypertrophic cardiomyopathy or dilated cardiomyopathy or infiltrative cardiomyopathy or constrictive cardiomyopathy
9. a history of congenital heart disease
10. a history of pulmonary hypertension
11. chronic atrial fibrillation or significant arrhythmia
12. a history of intracardiac device implantation
13. uncontrolled hypertension (systolic blood pressure > 160mm Hg or diastolic blood pressure > 100 mm Hg)
14. alanine Aminotransferase > 3 times upper limit)
15. acute infection
16. suspected or diagnosed with malignancy
17. a history of autoimmune disease
18. limited to or dependent on daily activities
19. life expectancy less than a year
20. Acute coronary syndrome or received a percutaneous coronary intervention or received a coronary artery graft bypass surgery or stroke within 3 months
21. Diabetes with insulin treatment or glucagon-like peptide 1 receptor agonist treatment
22. Anemia (hemoglobin < 11 mg/dl in mem or <10mg/dl in women)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of average E/e' | At day1 and at week 12
  the mean change of average E/e' in each group
Difference of average E/e' | At day1 and at week 12
  the mean difference of average E/e' between among three groups
Automate office blood pressure (AOBP) | At day1 and at week 12
  the mean difference of AOBP among three groups

SECONDARY OUTCOMES:
Change of xanthine oxidase activity | At day1 and at week 12
  the mean change of xanthine oxidase activity in each group
Difference of xanthine oxidase activity | At day1 and at week 12
  the mean difference of xanthine oxidase activity among three groups
Change of left ventricular mass index | At day1 and at week 12
  the mean change of left ventricular mass index in each group
Difference of left ventricular mass index | At day1 and at week 12
  the mean difference of left ventricular mass index among three groups
Change of tumor necrosis factor alpha | At day1 and at week 12
  the mean change of tumor necrosis factor alpha in each group
Difference of tumor necrosis factor alpha | At day1 and at week 12
  the mean difference of tumor necrosis factor alpha among three groups
Change of high-sensitivity interleukin-6 | At day1 and at week 12
  the mean change of high-sensitivity interleukin-6 in each group
Difference of high-sensitivity interleukin-6 | At day1 and at week 12
  the mean difference of high-sensitivity interleukin-6 among three groups
Change of thioredoxin | At day1 and at week 12
  the mean change of Thioredoxin in each group
Difference of Thioredoxin | At day1 and at week 12
  the mean difference of Thioredoxin among three group
Change of fibroblast growth factor 23 | At day1 and at week 12
  the mean Change of fibroblast growth factor 23 in each group
Difference of fibroblast growth factor 23 | At day1 and at week 12
  the mean difference of fibroblast growth factor 23 among three groups
Change of Dickkopf-related protein 3 | At day1 and at week 12
  the mean change of Dickkopf-related protein 3 in each group
Difference of Dickkopf-related protein 3 | At day1 and at week 12
  the mean difference of Dickkopf-related protein 3 among three groups
Change of galectin-3 | At day1 and at week 12
  the mean change of galectin-3 in each group
Difference of galectin-3 | At day1 and at week 12
  the mean difference of galectin-3 among three groups
Change of ST2 | At day1 and at week 12
  the mean change of ST2 in each group
Difference of ST2 | At day1 and at week 12
  the mean difference of ST2 among three groups

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Wei Liu, M.D., Principal Investigator — 1.Tri-service General hospital, Songshan branch, Taipei, Taiwan
Locations (1):
- Tri-service General Hospital, songshan branch, Taipei, Songshan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No